CLINICAL TRIAL: NCT06347588
Title: Novel HBV Biomarkers to Assess the Risk of Reactivation of Occult Hepatitis B in Cancer Patients During Immunotherapy: an Observational Prospective Multicenter Study.
Brief Title: Risk of Reactivation of Occult Hepatitis B in Cancer Patients During Immunotherapy.
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Angioletta Lasagna, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: OBI&ICI
Record Dates: First submitted 2024-03-26; First posted 2024-04-04 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Occult Hepatitis B Infection in Cancer Patients
MeSH Terms: interventions — Hepatitis B Surface Antigens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational: Blood sample of HVB-specific Elispot assay, HBSAg, HBV-DNA — Blood sample at baseline, week 4, month 3, 6, 9,12.

SUMMARY:
The goal of this observational study is to evalue the cumulative proportion of patients with OBI who do not develop HBsAg seroreversion and/or an increase of serum HBV DNA by at least 1 log above the lower limit of detection of the assay in a patient who had previously undetectable HBsAg and HBV DNA in serum during the study.

ELIGIBILITY:
Inclusion Criteria:

* Life-expectancy (as estimated by treating physician) ≥ 6 months;
* Patients HBsAg negative
* Patients HBcAb positive with or without HBV-DNA detectable
* Patients with cancer undergoing immunotherapy with or without chemotherapy

Exclusion Criteria:

* Patients who did not give informed consent
* Patients under prophylaxis for HBV
* Patients vaccinated for hepatitis B
* Patients with HBsAg positivity
* Patients with HIV positivity
* Patients with current history of alcohol (more than 5 alcohol unit daily) and drug use
* Patients with other cause of liver disease with known etiology (autoimmune liver disorder and storage liver disease)
* Patients with current active Hepatitis C virus (HCV-positive)
* Patients with hepatocellular carcinoma (HCC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors who have an occult hepatitis B infection and who need to start immunotherapy treatment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the cumulative proportion of patients with OBI who do not develop one seroreversion of HBsAg and/or an increase in serum HBV DNA of at least 1 log above the lower limit of detection of the test in a patient who had previously HBsAg and HBV | 3 weeks after first cycle of therapy and every 3 months until the end of the study
  Occult hepatitis B (OBI) detectable in serum HBV DNA, negative antigen test surface hepatitis B (HBsAg) and with positivity to anti-HBc (OBI seropositive).
  pOBI: Based on the intermittent detection of HBV DNA, we define pOBI (OBI potential) patients with negative HBV-DNA and positivity to anti-HBc.

SECONDARY OUTCOMES:
Evaluation of the incidence of reactivation in patients during immunotherapy | 3 weeks after first cycle of therapy and every 3 months until the end of the study
  Evaluation of the incidence of reactivation in patients during immunotherapy
Evaluation of the association between HBV-specific T-cell response and HBV reactivation | 3 weeks after first cycle of therapy and every 3 months until the end of the study
  Evaluation of the association between HBV-specific T-cell response and HBV reactivation
Analysis of the incidence of reactivation of HBV in patients with p-OBI according to tumor characteristics (histology and stage) and type and line of treatment (immunotherapy, combined treatment with chemotherapy + immunotherapy). | 3 weeks after first cycle of therapy and every 3 months until the end of the study
  Analysis of the incidence of reactivation of HBV in patients with p-OBI according to tumor

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Matteo Pavia, Pavia, PV, Italy